CLINICAL TRIAL: NCT00654524
Title: A Randomized Study Comparing Goserelin or Expectant Management Following Laparoscopic Surgery for Advanced Endometriosis
Brief Title: Randomized Study of Gonadotropin-releasing-hormone Agonist (GnRH-a) or Expectant Management for Endometriosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: XINMEI ZHANG, Women's Hospital School of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D8664L0001; ChiCTR-TRC-00000068
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2008-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; Recurrence; Pregnancy Rate; Laparoscopy; Gonadotropin-Releasing Hormone
MeSH Terms: conditions — Endometriosis; Recurrence | interventions — Gonadotropin-Releasing Hormone; Goserelin; Calcium Carbonate; tibolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in this arm will be treated with goserelin depot-3.6mg plus add-back therapy.
  Interventions: Drug: gonadotropin-releasing-hormone agonist (GnRHa) - Goserelin
- 2 (No Intervention): The patient with advanced endometriosis（stage III-IV）confirmed histologically after conservative laparoscopic surgery will be suggested to prepare for spontaneous pregnancy rather than any medical administration.

INTERVENTIONS:
Drug: gonadotropin-releasing-hormone agonist (GnRHa) - Goserelin — The patient will be managed with GnRH-a injection (Goserelin 3.6mg) every 4 weeks for 6 months plus add-back therapy (Caltrate With Vitamin D 600mg p.o. q.d.& Livial 1.25-2.5mg p.o. q.d.) if needed.
  Other Names: Goserelin; Caltrate With Vitamin D 600; Livial
  Arms: 1

SUMMARY:
The purpose of this study is to identify the recurrent rate and pregnancy rate of advanced endometriosis after laparoscopic surgery plus GnRHa goserelin acetate treatment.

DETAILED DESCRIPTION:
In order to decrease endometriosis recurrence and enhance pregnancy rate after surgical therapy, it has been proposed to use a post-surgical gonadotropin-releasing-hormone agonist (GnRHa) treatment. Data on the short-term recurrence of advanced endometriosis is rare. Although operative treatment has resulted in increasing pregnancy rate comparing non surgery management for moderate to severe endometriosis, very few data of spontaneous pregnancy rate are available comparing GnRHa treatment or expectant management after surgery treatment. In this situation, the investigators conduct a prospective, randomized, controlled study to determine whether postoperative GnRHa (goserelin acetate) therapy for advanced endometriosis is effective in reducing endometriosis recurrence rate and improving reproductive outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Normal menstruation for 3 months before enrollment (25-35 days）
* Advanced endometriosis confirmed histologically (r-AFS score III-IV) with laparoscopy or laparotomy-pelvic pain and/or dysmenorrhea and/or dyspareunia
* Agreement on the strict follow-up plan
* Without previous hormonal treatment
* Using nonhormonal method of contraception during this study

Exclusion Criteria:

* Serious heart diseases/pulmonary/liver/kidney diseases
* Previous non-endometriosis relevant surgery possibly influence to abdominal or pelvic pain
* Suspected malignancy in endometriosis
* Coagulation disorders with hemorrhagic tendency
* Pregnancy or lactation
* Allergy to GnRHa
* Previous ineffective treatment with GnRHa

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The recurrent rate of advanced endometriosis | within one year after surgery or GnRH-a management

SECONDARY OUTCOMES:
The pregnancy rate following laparoscopic surgery for advanced endometriosis | within one year after surgery or GnRH-a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xinmei Zhang, Prof., Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China